CLINICAL TRIAL: NCT05044572
Title: Comparison of Open Chain Kinetic Exercises and Forward Head Posture Correction on Scapular Symmetry and Glenohumeral Disability in Office Workers With Type II Scapular Dyskinesia
Brief Title: Comparison of Open Chain Kinetic Exercises and Forward Head Posture Correction in Type II Scapular Dyskinesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/0122 Sidra Ali
Record Dates: First submitted 2021-09-13; First posted 2021-09-16 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Dyskinesias
Keywords: Scapula
MeSH Terms: conditions — Dyskinesias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open chain kinetic exercises (Experimental)
  Interventions: Other: Open chain kinetic exercises
- Forward head posture correction exercises (Experimental)
  Interventions: Other: Forward head posture correction exercises

INTERVENTIONS:
Other: Open chain kinetic exercises — Group A will perform open chain kinetic exercises Before the intervention all the participants will perform 20 minutes of warm up and 10 minutes of cool down. The Open kinematic chain exercises(Three sets of each exercise while one set of each exercise will be performed at the setup and remaining two sets will be guided to the patient as a home plan)-:Blackburn exercises ( 20 repetitions ) , Dynamic hug( 10 repetitions), W exercise(10 repetitions), lunges with dumbbells-forward(10 repetitions with half kg dumbbell), upward and diagonal, and Pectoralis minor stretching(3 to 5 stretches)will be performed
  Arms: Open chain kinetic exercises
Other: Forward head posture correction exercises — PatienGroup B participants will perform forward head correction exercise(22) Chin tuck Patient will Stand with upper back against a wall, feet shoulder-width apart. • Face forward, tuck your chin down, and pull head back until it meets the wall. • t
  Arms: Forward head posture correction exercises

SUMMARY:
The objective of this study is to compare the effect of open chain kinetic exercises and forward head posture correction on scapular symmetry and glenohumeral disability in office workers with type II scapular dyskinesis.

DETAILED DESCRIPTION:
The scapula plays a crucial role in coordinating and maintaining complex shoulder kinematics. The rotator cuff (RC) and the scapula control energy and force transfer for glenohumeral (GH) and scapulothoracic (ST) movements. From a biomechanical perspective, the shoulder range of motion (ROM) covers almost 65% of a spherical joint whose stability is ensured by several factors such as bone integrity, muscle activity, and ligaments.The RC and scapula allow for three-dimensional movements of the shoulder by limiting excessive translations that may compromise the joint integrity.The overall prevalence of scapular dyskinesis was 90.08%, and the highest frequency was found at the resting position.

Association between ergonomic risk level and scapular dyskinesis in office workers in 2020. It was a cross sectional study A lateral scapular slide test (LSST) was used to evaluate scapular dyskinesis, and the quick exposure check (QEC) method was used to analyze the ergonomic risk level. results indicate that patients with scapular dyskinesis have a high ergonomic risk level.

A defective scapular posture, caused by muscular imbalances, also generates imbalances of length and muscular strength in the muscles, altering the mechanics of the glenohumeral joint. A forward bending of the scapula is associated with a retracted minor pectoral muscle and possibly anterior serratus weakness or trapezius. This scapular posture alters the humeral posture on the glenoid, assuming a relatively abducted and internally rotated position, resulting in retracted glenohumeral internal rotators and elongated or weak lateral rotators.

SW Christensen et al has stated in an article that the key group that might be related with scapular dyskinesis and work-related pain in office workers is the axioscapular muscles. These muscles attach between the scapula to the axis of the body consisted of serratus anterior, Pectoralis minor, rhomboids, levator scapulae and three parts of trapezius.

Study in 2016 in which the deeper lying (Levator Scapulae, Pectoralis Minor (Pm) and Rhomboid major) and superficial lying (Trapezius and Serratus Anterior) scapulothoracic muscles' activity was investigated with fine-wire and surface EMG, concluded that In the presence of idiopathic neck pain, higher Pectoralis minor activity during the towel wall slide was found. Patients with neck pain and scapular dyskinesis showed lower MT(middle trapezius) activity in comparison with healthy controls with scapular dyskinesis during scaption.

In 2018 The results showed high incidence of axioscapular muscle adaptations including of decreased flexibility of pectoralis minor, upper trapezius and levator scapulae in all subtypes as well as decreased performance of serratus anterior, middle trapezius, lower trapezius and rhomboids. The high incidence of postural deviations including forward head, rounded shoulder and thoracic hyper-kyphosis were also found in all subtypes of scapular dyskinesis. The participants were symptomatic office workers with different subtypes of scapular dyskinesis. They were evaluated the subtypes of scapular dyskinesis corresponded with flexibility of pectoralis minor, upper trapezius and levator scapulae using muscle length tests. The performances of serratus anterior, upper trapezius, middle trapezius, lower trapezius and rhomboids were also examined using manual muscle test. The postural deviations of cervical, shoulder and thoracic were also investigated using postural analysis methods.

Conventional therapeutic exercise programs are commonly used to treat patients with scapular dyskinesis. It is common for physical therapists to treat patients with shoulder pain and scapular dyskinesis. Treatment techniques to address dyskinesis include manual neuromuscular facilitation, tactile cueing, visual feedback, electrical stimulation, supervised exercise, mobilization, strengthening, electromyography, and other interventions.

An RCT in which eleven asymptomatic university students representing 15 scapulae with a positive Scapular Dyskinesis Test were recruited as subjects. Participants were randomized into exercise and electrical stimulation (ESTherex) or exercise and sham electrical stimulation (ShamTherex) and stated that Electrical stimulation with exercises for scapular dyskinesis showed improvements in spine to scapula distance at 120 degrees of shoulder abduction.

The literature has proved that shoulder stabilization training strengthens the scapular muscles, closed chain and open chain kinetic exercises are also beneficial thereby resolving the SD. But as FHP can lead to SD, among the correction of FHP or open chain kinetic exercises which one is more effective to treat SD type II it has not been compared before. There is also paucity of literature available on open chain kinetic exercises and forward head posture correction exercises on scapular symmetry and glenohumeral disability in office workers with type II scapular dyskinesis. Hence this study aims to compare the effect of open chain kinetic exercises and forward head posture correction on scapular symmetry and glenohumeral disability in office workers with type II Scapular dyskinesis.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female office workers
* In the age group of 20 to 40 years
* With at least one year work experience
* Individuals with Type II scapular dyskinesia (1-1.5 cm dif¬ference)
* Individuals with forward head posture

Exclusion Criteria:

* Any Congenital abnormality
* Neurological deficit
* Received physiotherapy treatment in past three months

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
SPADI questionnaire | 4 week
  The Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability.
Lateral Scapular Slide Test (LSST) | 4 weeks
  Lateral Scapular Slide Test (LSST) will be used to evaluate the scapular dyskinesis. LSST asses scapular asymmetry under varying load positions. Measurements of scapular position are taken while scapular position with the arm abducted 0, 45, and 90 degrees in the coronal plane. Distance from the inferior angle of the scapula to the spinous process of the thoracic vertebra in the same horizontal plane was measured in all 3 position .If the distance is greater than 1.5 cm, it means LSST is positive
Forward head posture measurement using Image J software | 4 weeks
  Forward head posture measurement will be assessed using a digitized , lateral view photograph(Sony 16.1 M pixels camera ) of the subject in his or her usual standing posture. The tragus of the subject's ear will be marked and a reflexive marker will be attached to the skin overlying C7 vertebrae. Once the photograph obtained we will use ImageJ software (20)to measure FHP quantified by the craniovertebral angle (The angle between the horizontal line passing through the C7 and a line extending from tragus of ear to C7). An angle less than 50-53 degrees may indicate FHP . Thereby, the smaller the CV angle, the greater the disability.
Universal Goniometer | 4 weeks
  In Type 2 Scapula Dyskinesia, weakness of the serratus anterior results in reduction in both glenohumeral flexion and abduction .So these ranges will be measured before and after intervention in both groups with the help of goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Saima Zahid, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Sarwat Anwar Medical Complex Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lefevre-Colau MM, Nguyen C, Palazzo C, Srour F, Paris G, Vuillemin V, Poiraudeau S, Roby-Brami A, Roren A. Recent advances in kinematics of the shoulder complex in healthy people. Ann Phys Rehabil Med. 2018 Jan;61(1):56-59. doi: 10.1016/j.rehab.2017.09.001. Epub 2017 Sep 28. No abstract available. PMID 28964876
- [Background] Lefevre-Colau MM, Nguyen C, Palazzo C, Srour F, Paris G, Vuillemin V, Poiraudeau S, Roby-Brami A, Roren A. Kinematic patterns in normal and degenerative shoulders. Part II: Review of 3-D scapular kinematic patterns in patients with shoulder pain, and clinical implications. Ann Phys Rehabil Med. 2018 Jan;61(1):46-53. doi: 10.1016/j.rehab.2017.09.002. Epub 2017 Oct 5. PMID 28987866
- [Background] Kibler WB, Sciascia A. The role of the scapula in preventing and treating shoulder instability. Knee Surg Sports Traumatol Arthrosc. 2016 Feb;24(2):390-7. doi: 10.1007/s00167-015-3736-z. Epub 2015 Aug 1. PMID 26231154
- [Background] Deng S, Chen K, Ma Y, Chen J, Huang M. The Influence of Test Positions on Clinical Assessment for Scapular Dyskinesis. PM R. 2017 Aug;9(8):761-766. doi: 10.1016/j.pmrj.2016.11.011. Epub 2016 Dec 1. PMID 27916706
- [Background] Panagiotopoulos AC, Crowther IM. Scapular Dyskinesia, the forgotten culprit of shoulder pain and how to rehabilitate. SICOT J. 2019;5:29. doi: 10.1051/sicotj/2019029. Epub 2019 Aug 20. PMID 31430250
- [Background] Longo UG, Risi Ambrogioni L, Berton A, Candela V, Massaroni C, Carnevale A, Stelitano G, Schena E, Nazarian A, DeAngelis J, Denaro V. Erratum: Longo, U.G., et al. Scapular Dyskinesis: From Basic Science to Ultimate Treatment. International Journal of Environmental Research and Public Health 2020, 17(8), 2974. Int J Environ Res Public Health. 2020 May 27;17(11):3810. doi: 10.3390/ijerph17113810. PMID 32471164
- [Background] Singla D, Veqar Z. Association Between Forward Head, Rounded Shoulders, and Increased Thoracic Kyphosis: A Review of the Literature. J Chiropr Med. 2017 Sep;16(3):220-229. doi: 10.1016/j.jcm.2017.03.004. Epub 2017 Sep 28. PMID 29097952
- [Background] Ozdemir F, Toy S. Evaluation of scapular dyskinesis and ergonomic risk level in office workers. Int J Occup Saf Ergon. 2021 Dec;27(4):1193-1198. doi: 10.1080/10803548.2020.1757307. Epub 2020 Jun 22. PMID 32306852
- [Background] Christensen SW, Hirata RP, Graven-Nielsen T. The effect of experimental neck pain on pressure pain sensitivity and axioscapular motor control. J Pain. 2015 Apr;16(4):367-79. doi: 10.1016/j.jpain.2015.01.008. Epub 2015 Jan 29. PMID 25640292
- [Background] Castelein B, Cools A, Parlevliet T, Cagnie B. Are chronic neck pain, scapular dyskinesis and altered scapulothoracic muscle activity interrelated?: A case-control study with surface and fine-wire EMG. J Electromyogr Kinesiol. 2016 Dec;31:136-143. doi: 10.1016/j.jelekin.2016.10.008. Epub 2016 Oct 19. PMID 27816845